CLINICAL TRIAL: NCT00680498
Title: Combination Lucentis and Ocular Photodynamic Therapy With Visudyne, With Evaluation-based Retreatment
Acronym: CLOVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Illinois Retina Associates (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clover 1
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Ranibizumab; Lucentis; Photodynamic Therapy; Verteporfin; Visudyne
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Photochemotherapy; Verteporfin

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ranibizumab
- 2 (Active Comparator)
  Interventions: Drug: Ranibizumab plus Photodynamic therapy

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5 mg
  Other Names: Lucentis
  Arms: 1
Drug: Ranibizumab plus Photodynamic therapy — Ranibizumab 0.5mg, combined with photodynamic therapy with Verteporfin (dosage per label)
  Other Names: Lucentis; Visudyne
  Arms: 2

SUMMARY:
This is a one-year, randomized, single-center open-label pilot study of the safety and efficacy of combination ranibizumab and PDT for AMD. Eligible subjects will be randomized to either combination treatment, or ranibizumab monotherapy (control group).

The combination treatment group will receive ranibizumab, followed 1 week later by verteporfin PDT. Additional treatments will be based on evidence of active disease (subretinal fluid on OCT or leakage on FA): repeat ranibizumab injections will be allowed monthly, and repeat PDT will be allowed every 3 months.

The control group will receive "standard-of-care" ranibizumab monotherapy according to the protocol currently followed by most retinal specialists. Ranibizumab injections will be given at baseline and months one and two. Additional injections will be given at each monthly visit at which there is evidence of active disease by visual acuity, OCT and FA criteria.

ELIGIBILITY:
Inclusion Criteria:

* Presence of subfoveal CNV due to AMD, less than 9 disc areas in extent
* Vision 20/40 to 20/800 Snellen equivalent
* Age > 50 years
* Ability to provide written informed consent and comply with study assessments for the full duration of the study

Exclusion Criteria:

* Intraocular surgery or injection within 30 days prior to enrollment in the study eye
* Intravitreal triamcinolone within the past 6 months in the study eye
* History of prior PDT treatment in the study eye
* History of argon laser treatment of subfoveal CNV in the study eye
* Other vision-limiting disease (e.g. advanced glaucoma, prior vascular occlusion, dense amblyopia) in the study eye
* Clinically significant intraocular inflammation in the study eye
* No light perception in the fellow eye
* Anterior segment opacity preventing adequate visualization of fundus for FA or OCT
* Are currently participating in another clinical trial
* Women of childbearing potential not using adequate contraception, as well as women who are breastfeeding
* Known sensitivity to study drug(s) or class of study drug(s)
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine whether combination treatment can maintain or improve visual acuity within 3 lines of baseline visual acuity. | 1 year

SECONDARY OUTCOMES:
Determination of whether combination treatment can minimize the number of re-treatments required to stabilize vision. | 1 year
Determination of change in visual acuity from baseline. | 1 year
Determination of change in retinal thickness by optical coherence tomography (OCT). | 1 year
Determination of change in angiographic leakage from CNV. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pauline T Merrill, MD, Principal Investigator — Illinois Retina Associates
Locations (1):
- Illinois Retina Associates, Oak Park, Illinois, United States